CLINICAL TRIAL: NCT01145755
Title: A Phase IIa, Multi-centre, Randomized, Double-Blind, Double-Dummy, Active and Placebo Controlled, Parallel Group Study to Assess the Effectiveness and Safety of AZD2066 After 6 Weeks of Treatment in Patients With Major Depressive Disorder - D0475C00020
Brief Title: 6-week Study Treatment to Evaluate the Safety and Effectiveness of AZD2066 in Patients With Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0475C00020
Record Dates: First submitted 2010-05-27; First posted 2010-06-17 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — AZD2066; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- AZD2066 (Experimental)
  Interventions: Drug: AZD2066
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Duloxetine (Active Comparator): Duloxetine
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: AZD2066 — 18 mg once daily
  Arms: AZD2066
Drug: Placebo
  Arms: Placebo
Drug: Duloxetine — 60 mg once daily
  Arms: Duloxetine

SUMMARY:
This is a 6-week study treatment to evaluate the safety and effectiveness of AZD2066 in patients with major depressive disorder.

DETAILED DESCRIPTION:
A Phase IIa, Multi-centre, Randomized, Double-Blind, Double-Dummy, Active and Placebo Controlled, parallel Group Study to Assess the Efficacy and Safety of AZD2066 after 6 weeks of treatment in Patients with Major Depressive Disorder - D0475C00020.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written, and dated Informed Consent
* Documented primary clinical diagnosis of Major Depressive Disorder

Exclusion Criteria:

* Patients with a secondary psychiatric disorder including bipolar disorder, psychotic disorders (i.e. schizophrenia, schizoaffective disorder, depression with psychotic features), GAD and social anxiety disorder
* Patients whose current episode of depression started less than 4 weeks before enrollment
* History of inadequate response of antidepressants during current depressive episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Malamut, Study Chair — AstraZeneca; Lora McGill, Principal Investigator — CNS Healthcare
Locations (13):
- United States (13):
  - Research Site, Garden Grove, California
  - Research Site, San Diego, California
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Rockville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Cedarhurst, New York
  - Research Site, Rochester, New York
  - Research Site, Portland, Oregon
  - Research Site, Memphis, Tennessee
  - Research Site, Friendswood, Texas
  - Research Site, Bellevue, Washington
  - Research Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted only in the United States (US). A total of 13 study centers enrolled 249 patients. First subject enrolled: 27 May 2010 Last subject last visit: 10 November 2010
Pre-assignment Details: Patients with major depressive disorder were included.
Groups:
- AZD2066: AZD2066 12 mg, 18 mg
- Duloxetine: Duloxetine 30 mg, 60 mg
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD2066 | Duloxetine | Placebo
Started | 40 | 47 | 44
Completed | 20 | 19 | 19
Not Completed | 20 | 28 | 25
Not completed — Adverse Event | 2 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Protocol Violation | 0 | 3 | 1
Not completed — Study Closure | 14 | 14 | 17
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Patient could not swollow medication | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Positive urine ethanol | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2066 | Duloxetine | Placebo | Total
Number analyzed (Participants) | 40 | 47 | 44 | 131
Age Continuous [Mean (Full Range); unit: Years] | 42.2 [21 to 60] | 39.9 [19 to 60] | 38.4 [20 to 61] | 40.1 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 30 | 77
  Male | 17 | 23 | 14 | 54

OUTCOME MEASURES:

1. Primary Outcome: MADRS Total Score Change From Baseline to Week 6
Description: Montgomery-Asberg Depression Rating Scale (MADRS): The MADRS is a 10-item scale for the evaluation of depressive symptoms (Montgomery et al 1979). Each MADRS item is rated on a 0 to 6 scale. Total score range from 0-60, where higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: scores on the scale
Arm/Group | AZD2066 | Duloxetine | Placebo
Number analyzed (Participants) | 39 | 45 | 40
scores on the scale | -13.1658 (2.11) [NA to NA] | -14.0271 (1.97) [NA to NA] | -14.1575 (2.16) [NA to NA]

2. Secondary Outcome: MADRS Response
Description: A MADRS responder at week 6 is defined as a patient with a reduction of at least 50% from baseline MADRS total score.
Time Frame: 6 weeks
Measure: Number; unit: Participants
Arm/Group | AZD2066 | Duloxetine | Placebo
Number analyzed (Participants) | 21 | 20 | 19
Participants | 9 | 9 | 9

3. Secondary Outcome: MADRS Remission
Description: A patient will be classified as in remission if their MADRS total score is ≤10 at Week 6
Time Frame: 6 weeks
Measure: Number; unit: Participants
Arm/Group | AZD2066 | Duloxetine | Placebo
Number analyzed (Participants) | 21 | 20 | 19
Participants | 5 | 8 | 7

ADVERSE EVENTS:
Arm/Group | AZD2066 | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/47 | 0/44
Other Adverse Events (participants affected / at risk) | 21/40 | 30/47 | 16/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2066 (N=40) | Duloxetine (N=47) | Placebo (N=44)
Ovarian mass (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2066 (N=40) | Duloxetine (N=47) | Placebo (N=44)
NAUSEA (Gastrointestinal disorders) | 6 | 12 | 4
DIARRHOEA (Gastrointestinal disorders) | 3 | 10 | 4
DRY MOUTH (Gastrointestinal disorders) | 1 | 7 | 4
CONSTIPATION (Gastrointestinal disorders) | 4 | 1 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0 | 0
IRRITABILITY (General disorders) | 2 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 3 | 1
INCREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 1
HEADACHE (Nervous system disorders) | 10 | 7 | 0
SOMNOLENCE (Nervous system disorders) | 2 | 5 | 0
DIZZINESS (Nervous system disorders) | 3 | 3 | 2
INSOMNIA (Psychiatric disorders) | 4 | 2 | 0
ANXIETY (Psychiatric disorders) | 2 | 0 | 2
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 5 | 1
RASH (Skin and subcutaneous tissue disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or presentation of results until the earlier of 1) the date of the first study results publication or 2) 18 months after completion or termination of the study.

AZ review 60 days prior submission and AZ has the possibility to further delay publication for an additional 90 days